CLINICAL TRIAL: NCT05029388
Title: Effects of Aerobic Exercise and High-Intensity Interval Training on the Mental Health of Adolescents Living in Poverty
Brief Title: Aerobic Exercise and High-Intensity Interval Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Education University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EdUHK
Record Dates: First submitted 2021-08-16; First posted 2021-08-31 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Mental Health
Keywords: adolescents; mental health; exercise; socioeconomic status; intervention
MeSH Terms: conditions — Psychological Well-Being; Motor Activity | interventions — Exercise; High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A total of 78 participants with low SES who are aged between 12 and 15 and studying in secondary one to three from local secondary schools will be recruited for this study. They will be randomly assigned to either an aerobic exercise group, an HIIT group, or a no-exercise control group. Participants in the first two groups will partake in a 10-week training program period, which will be conducted thrice a week on non-consecutive days.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Aerobic Exercise (Experimental): This experimental group will receive aerobic exericse. This group will be led by a certified personal trainer with at least three years of experience in guiding adolescents in group exercises. The aerobic exercise training will be conducted in the fitness room of a local sports center that is hosted by the Leisure and Cultural Services Department in Hong Kong.
  Interventions: Other: Aerobic Exercise
- High Intensity Interval Training (Experimental): This experimental group will receive high intensity interval training. This group will be led by a certified personal trainer with at least three years of experience in guiding adolescents in group exercises. The HIIT training will be conducted in the fitness room of a local sports center that is hosted by the Leisure and Cultural Services Department in Hong Kong.
  Interventions: Other: High Intensity Interval Training
- Control Group (No Intervention): This group will not take part in aerobic exercise and HIIT training programme. Participants will be given an exercise diary or logbook to keep track of their exercise habits (i.e., record the type of exercise/activity, hours, and intensity of exercise/activity every day) throughout the intervention periods.

INTERVENTIONS:
Other: Aerobic Exercise — The participants will complete three training sessions per week over 10 weeks. The aerobic training program will last for one hour. The session will include a 10-minute warm-up period, followed by a 45-minute aerobic workout, wherein the participants can choose to use either a treadmill, a cycle ergometer, or a rowing ergometer. After the workout, a five-minute period of stretching will be provided for cooling down. The intensity during the workout will be set at 40%-55% of the individual's maximum heart rate.
  Arms: Aerobic Exercise
Other: High Intensity Interval Training — The intervention will be conducted over a period of 10 weeks, while the participants will complete three training sessions per week. The HIIT training program will last for 30 minutes. The session will include a 10-minute warm-up period, followed by a 15-minute HIIT workout, and a 5-minute period of stretching to cool down. The exercises will include repeated, high-intensity intermittent bursts of vigorous activity at maximal effort. The HIIT will mainly include bodyweight exercises (e.g., push-ups, squats, lunges) that disregards equipment usage. The intensity during the workout will be set to 85%-95% of the individual's maximum heart rate. A half-day training workshop will be provided to the personal trainer to ensure that he/she knows the exercises and can demonstrate them to the participants.
  Arms: High Intensity Interval Training

SUMMARY:
The increasing rate of mental health issues among adolescents has recently been a considerable concern in Hong Kong. In particular, adolescents with low socioeconomic status (SES) are likely to experience poor mental health including low self-esteem and high levels of anxiety, anger, and depression. Previous research has found that physical activities have a positive impact on improving mental health outcomes among adolescents. However, approximately 96% of adolescents in Hong Kong fail to engage in regular exercises, which potentially increase risk of poor mental health. This study aims to (1) examine whether changes in the three indicators (reduced ill-being, enhanced well-being and cognitive functions) of mental health among adolescents with low socioeconomic status are evident before and after exercises. In addition, this study (2) compares the effectiveness of aerobic exercise and high-intensity interval training in these indicators among adolescents with low SES. A range of neuropsychological tests and psychometric scales will be used to measure the executive functions and indicators of psychological well-being and ill-being, which include enjoyment, self-efficacy, mood, depression, anxiety, and stress. It is hoped that the findings will help inform policymakers and practitioners for promoting the importance of physical exercises to enhance mental health.

DETAILED DESCRIPTION:
Adolescents' poor mental health provides serious implications for adult morbidity and mortality. Mental health involves the absence of mental illness and life satisfaction. In Hong Kong (HK), the mental health of adolescents has been a subject of considerable concern in recent years. A recent survey of 11,493 local citizens revealed that approximately 74% of adolescents below the age of 25 years exhibit moderate to high levels of depressive symptoms (e.g., depression, anxiety, and stress), 41% suffer moderate to high levels of post-traumatic stress symptoms, and 36% have both diagnoses. Previous research has also demonstrated that poor mental health is unevenly distributed across different socioeconomic groups and is highly clustered in families with socioeconomic status (SES).

Families with low SES are more deprived in multiple ways and suffer from numerous stressors related to finances, social relations, employment opportunities, and physical illness than families from other socioeconomic groups. For instance, adolescents with low SES often have worse access to education and social participation than their peers with an average or high SES. In addition, the results from a meta-analysis study of 34 countries from 2002 to 2010 indicated that adolescents with low SES are affected by physical symptoms and have poor mental health, including low self-esteem and high levels of anxiety, anger, and depression.

Physical exercise is presently considered as an effective intervention for its safe, nonpharmacological, and cost-effective nature that can provide a range of health benefits, including improvements in body composition and physical capacity, among individuals. Recent evidence has confirmed that physical exercise provides a positive effect on mental health outcomes for youth through physiological and psychological pathways.

Studies that are focused on physiological evidence have commonly demonstrated a direct positive effect of physical exercise on the individuals' neurological processes, thereby indicating that cardio activities are directly and immediately beneficial to mental health. Two main research streams that cite physiological evidence, namely, those that focus on monoamines and those that focus on endorphins are present. The first research stream reveals that physical activity upregulates the synaptic transmission of monoamines, including the three major neurotransmitters, namely, norepinephrine, dopamine, and serotonin. A similar effect has been found for antidepressant drugs, while exercise has been proven as effective as antidepressants for alleviating depressive symptoms among patients with major depression. The hypothesis regarding endorphin is also popular for explaining the impacts of aerobic exercise on mental health. Several researchers have believed that endorphins may lead to energy conservation during exercise and consequently exhibits psychological effects such as improved mood states and reduced anxiety. Direct evidence stating that physical activity can elevate the plasma endorphin levels also exists.

Although physiological evidence has established a direct association between physical activity and mental health, researchers are also keen to identify how physical activities may benefit mental health. Several researchers have conducted studies based on the three indicators of mental health that were proposed by Costigan et al. (2016), namely, (1) cognitive function, (2) well-being (e.g., enjoyment), and (3) ill-being (e.g., depression, negative affect).

With regard to cognitive function, a growing evidence indicates that participating in exercise positively affects the executive functions. Executive function is an umbrella term, which covers a wide array of cognitive processes that govern goal-directed actions and adaptive responses to novel, complex, or ambiguous situations. Numerous studies have found that intense physical exercise improves working memory inhibitory control, and cognitive flexibility in typical and low-income adolescents.

Physical exercise has been associated with improved well-being, including life satisfaction and self-esteem. Exercise is a challenging activity, but the process of engaging in exercise could provide individuals with a meaningful experience of mastery that may lead to improved mood states and self-confidence. Affect regulation theory suggests that exercise could regulate affect by reducing negative mood states and enhancing positive mood states conducive to mental well-being. Furthermore, as described in relevant literature, exercise could divert an individual from unfavourable stimuli (e.g., worries, stress, and depressive thoughts) leading to improved moods.

Physical exercise has also been associated with reduced ill-being. A meta-analysis of 73 studies confirmed that increased levels of physical activity exhibit significant effects on reducing depression, anxiety, psychological distress, and emotional disturbance among children Archer and Garcia (2017) found that regular physical exercise ameliorated the symptoms of anxiety and depression. Behavioral activation theory posits that depressive symptoms may be alleviated when individuals replaced passive activities with exercise and other entertaining activities.

Although a lack of consensus regarding the most effective training regimen for physical exercise is evident in clinical review studies from 2000 to 2014, Ranjbar et al. (2015) recommended the following components of an effective exercise program to benefit adolescents with poor mental health. Based on the frequency, intensity, time, and type (FITT) principle, an exercise program should include the characteristics, namely, (1) structured aerobic exercise, which requires the heart to pump oxygenated for delivering oxygen to working muscles and stimulates an increase in the heart rate (HR) and breathing rate; (2) group exercise, particularly for adolescents; (3) low (40%-55% VO2max) to moderate (65%-75% VO2max) intensity; (4) 45 to 60 minutes length of session; (5) frequency of at least three to four times per week, which is equal to 150 or above minutes of exercise per week; and (6) a duration equal to 10 weeks or above.

Overall, the extensive research has confirmed that physical exercise can significantly improve physical and mental health, while aerobic exercise has been the main focus of most previous studies. Research has recently been attempted to determine whether low-volume HIIT could be a time-efficient exercise strategy for improving health and fitness among the general population.

HIIT is a time-efficient type of aerobic training that involves a short duration of full-effort exercise, followed by a rest period. HIIT is mainly appealing because it can be completed in a relatively short period that results in equivalent physiological adaptations of long sessions of traditional aerobic training and improvements in physical and mental health. This strategy may be feasible and effective for increasing physical health outcomes among young people. Compared with low-intensity, high-volume (duration) endurance aerobic training (i.e., cycling), HIIT can result in better oxygen uptake, greater muscle deoxygenation, and better exercise performance. A previous study also revealed that patients participating in high-intensity interval running reported higher perceived enjoyment than those participating in moderate-intensity continuous running. A pilot study of a 10-week HIIT program resulted in improved metabolic outcomes among patients with schizophrenia, thereby supporting the benefits of HIIT for physical fitness and mental health. Further studies have also shown that HIIT reduces distress and anxiety.

Despite the promising evidence that supports the adoption of HIIT among adults with various conditions, limited research that targets adolescents, particularly those with low SES, is available. High-intensity activities performed in short, repeated bouts with periods of recovery in-between could be an achievable and enjoyable alternative to high-volume continuous exercise for adolescents, including "low-active" adolescents.

The conditions and ability of poor individuals to manage and potentially escape from poverty are the core of policy agendas and the ethical and economic concerns among societies. Behavioral research has recently been applied to policy-relevant challenges and has explored the significant potential of simple interventions to influence cognition and behavior. Poor individuals, particularly young poor individuals in HK, have received little attention as part of this endeavour despite their characteristics that satisfy the qualifications of clear candidates for interventions that could improve disadvantaged situations.

Although several longitudinal studies have confirmed that growing up in a disadvantaged family is a significant risk factor of poor mental health, numerous research gaps should be addressed by further investigation. For instance, most studies on mental health and socioeconomically disadvantaged adolescents have been restricted to understanding and confirming the link between mental health and SES. Research that aims to examine whether mental health could be enhanced through physical exercise is scarce. However, such research would be extremely meaningful for expanding early interventions. To date, a steady decline in the number of physically active students in HK is evident. Furthermore, the situation among adolescents in HK is worse given that 96% of them are insufficiently active. Hence, a considerable need for this kind of research arises to arouse public awareness on the link between physical activity and mental health. Although previous studies have reported the improvements in the mental health of adolescents after exercise sessions, a lack of follow-up data is available on assessing the sustainability of the exercise intervention with moderate intensity under long duration. In addition, relatively few studies directly compared the effects of aerobic exercise and HIIT on the mental health of adolescents with low SES. Given that HIIT training has become popular and effective on improving health and well-being, HIIT exercise should be used as the comparison group to examine the effectiveness of traditional aerobic exercise.

Following the health benefits of regular exercise and the limited research on exercise-based interventions (aerobic exercise vs. HIIT) with low-SES adolescents, this study primarily aims to investigate the effectiveness of aerobic exercise and HIIT on the three indicators of mental health among low-SES adolescents. This paper particularly intends to answer two research questions, namely, (1) Is there any change in the three indicators of mental health (i.e., cognitive function, well-being, and ill-being) before and after exercise? (2) Which exercise regimen (aerobic exercise or HIIT) is more effective in reducing ill-being and enhancing well-being and cognitive function among adolescents with low SES?

ELIGIBILITY:
Inclusion Criteria:

* Studying in secondary grades one to three
* Between 12 and 15 years old
* Belongs to a family with a household income below half of the median household income reported in HK, which was adjusted by household size

Exclusion Criteria:

* Hypertension or diabetes mellitus without control
* A history of brain injury and other neurological disease, epilepsy, or myocardial infarction
* Musculoskeletal disease
* Use medication that affects heart rate (e.g., beta-blockers, asthma medications, stimulants, digoxin, antiarrhythmic agents)
* Cardiovascular disease

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 78 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Physical Activity Enjoyment Scale (S-PACES) | One week before pretest
  This scale will be utilized to measure enjoyment. The S-PACES includes seven negatively worded items (e.g., "It is not at all interesting"), anchored on a five-point Likert scale that ranges from 1 (disagree a lot) to 5 (agree a lot).
Physical Activity Enjoyment Scale (S-PACES) | 10 weeks after intervention
  This scale will be utilized to measure enjoyment. The S-PACES includes seven negatively worded items (e.g., "It is not at all interesting"), anchored on a five-point Likert scale that ranges from 1 (disagree a lot) to 5 (agree a lot).
Physical Activity Enjoyment Scale (S-PACES) | 3 months after intervention
  This scale will be utilized to measure enjoyment. The S-PACES includes seven negatively worded items (e.g., "It is not at all interesting"), anchored on a five-point Likert scale that ranges from 1 (disagree a lot) to 5 (agree a lot).
General Self-Efficacy Scale (GSES) | One week before pretest
  This scale will be administered to measure the adolescents' self-efficacy. The GSES contains 10 items (e.g., "I can constantly manage to solve difficult problems if I try hard enough"), with responses ranging from 1 (not at all true) to 4 (exactly true).
General Self-Efficacy Scale (GSES) | 10 weeks after intervention
  This scale will be administered to measure the adolescents' self-efficacy. The GSES contains 10 items (e.g., "I can constantly manage to solve difficult problems if I try hard enough"), with responses ranging from 1 (not at all true) to 4 (exactly true).
General Self-Efficacy Scale (GSES) | 3 months after intervention
  This scale will be administered to measure the adolescents' self-efficacy. The GSES contains 10 items (e.g., "I can constantly manage to solve difficult problems if I try hard enough"), with responses ranging from 1 (not at all true) to 4 (exactly true).
Satisfaction with Life Scale (SWLS) | One week before pretest
  The scale will be used to measure life satisfaction. This scale is a short five-item (e.g., "I am satisfied with my life") scale based on a seven-point rating scale that ranges from 1 (strongly disagree) to 7 (strongly agree).
Satisfaction with Life Scale (SWLS) | 10 weeks after intervention
  The scale will be used to measure life satisfaction. This scale is a short five-item (e.g., "I am satisfied with my life") scale based on a seven-point rating scale that ranges from 1 (strongly disagree) to 7 (strongly agree).
Satisfaction with Life Scale (SWLS) | 3 months after intervention
  The scale will be used to measure life satisfaction. This scale is a short five-item (e.g., "I am satisfied with my life") scale based on a seven-point rating scale that ranges from 1 (strongly disagree) to 7 (strongly agree).
21-item Depression Anxiety Stress Scale (DASS-21) | One week before pretest
  The DASS-21 scale will be used to measure depression (e.g., "I felt that I lack something to look forward to"), anxiety (e.g., "I felt that I was close to panic"), and stress (e.g., "I found it difficult to relax") among adolescents. The respondents will be asked to rate the items through a four-point combined severity/frequency scale that ranges from 0 (not applicable to me at all) to 3 (extremely applicable to me) based on their experiences that are related to each item over the past week.
21-item Depression Anxiety Stress Scale (DASS-21) | 10 weeks after intervention
  The DASS-21 scale will be used to measure depression (e.g., "I felt that I lack something to look forward to"), anxiety (e.g., "I felt that I was close to panic"), and stress (e.g., "I found it difficult to relax") among adolescents. The respondents will be asked to rate the items through a four-point combined severity/frequency scale that ranges from 0 (not applicable to me at all) to 3 (extremely applicable to me) based on their experiences that are related to each item over the past week.
21-item Depression Anxiety Stress Scale (DASS-21) | 3 months after intervention
  The DASS-21 scale will be used to measure depression (e.g., "I felt that I lack something to look forward to"), anxiety (e.g., "I felt that I was close to panic"), and stress (e.g., "I found it difficult to relax") among adolescents. The respondents will be asked to rate the items through a four-point combined severity/frequency scale that ranges from 0 (not applicable to me at all) to 3 (extremely applicable to me) based on their experiences that are related to each item over the past week.
Brunel Mood Scale (BRUMS-C) | One week before pretest
  The BRUMS-C will be created based on the work of Terry, Lane, Lane, and Keohane (1999) to assess the mood among Chinese students and adults. The BRUMS-C is a 23-item inventory with five negative mood dimensions, namely, anger, confusion, depression, fatigue, and tension. Respondents will be asked to indicate their feelings (e.g., angry, unhappy, or nervous) through a five-point Likert scale that ranges from 0 (not at all) to 4 (extremely).
Brunel Mood Scale (BRUMS-C) | 10 weeks after intervention
  The BRUMS-C will be created based on the work of Terry, Lane, Lane, and Keohane (1999) to assess the mood among Chinese students and adults. The BRUMS-C is a 23-item inventory with five negative mood dimensions, namely, anger, confusion, depression, fatigue, and tension. Respondents will be asked to indicate their feelings (e.g., angry, unhappy, or nervous) through a five-point Likert scale that ranges from 0 (not at all) to 4 (extremely).
Brunel Mood Scale (BRUMS-C) | 3 months after intervention
  The BRUMS-C will be created based on the work of Terry, Lane, Lane, and Keohane (1999) to assess the mood among Chinese students and adults. The BRUMS-C is a 23-item inventory with five negative mood dimensions, namely, anger, confusion, depression, fatigue, and tension. Respondents will be asked to indicate their feelings (e.g., angry, unhappy, or nervous) through a five-point Likert scale that ranges from 0 (not at all) to 4 (extremely).
Blood Pressure | Resting state at baseline
  Blood pressure will be measured with an automated blood pressure monitoring device. The participants will be given 10-minute rest before the measurement. The systolic and diastolic blood pressure will be measured thrice, with a one-minute interval between readings. If the blood pressure differed by more than 5 mm Hg, then additional readings will be obtained. A mean of the three consecutive readings will be used as the examination value. The unit of measurement for blood pressure is mmHg.
Blood Pressure | At the end of training
  Blood pressure will be measured with an automated blood pressure monitoring device. The participants will be given 10-minute rest before the measurement. The systolic and diastolic blood pressure will be measured thrice, with a one-minute interval between readings. If the blood pressure differed by more than 5 mm Hg, then additional readings will be obtained. A mean of the three consecutive readings will be used as the examination value. The unit of measurement for blood pressure is mmHg.
Resting Heart Rate | Resting state at baseline
  The resting heart rate will be measured through a wireless heart rate monitor that will be worn by the participants (Polar Electro OY, Finland) for one minute after their 10-minute rest. The unit of measurement for heart rate is bpm (beats per minute).
Resting Heart Rate | At the end of training
  The resting heart rate will be measured through a wireless heart rate monitor that will be worn by the participants (Polar Electro OY, Finland) for one minute after their 10-minute rest. The unit of measurement for heart rate is bpm (beats per minute).
Body Mass Index | Resting state at baseline
  The body weight and height will be measured using an electronic digital scale and a stadiometer, respectively. The body mass index (BMI) will be calculated by dividing body weight (kg) by height (m^2).
Body Mass Index | At the end of training
  The body weight and height will be measured using an electronic digital scale and a stadiometer, respectively. The body mass index (BMI) will be calculated by dividing body weight (kg) by height (m^2).
Waist-to-Hip Ratio | Resting state at baseline
  The waist circumference and hip circumference will be measured twice using an anthropometric tape while the participants stand erect and relaxed with their arms at their sides and feet positioned close together. The waist circumference will be measured between the upper border of the iliac crest and the lowest border of the rib cage at the end of normal expiration. The hip circumference will be measured at the widest part of the hip at the level of the greatest trochanter. The tape will be positioned at a level that is parallel to the floor. The unit of measure will be in centimeters (cm) to the nearest 0.1 cm. The waist-to-hip ratio will be calculated as the ratio of the waist-to-hip circumference.
Waist-to-Hip Ratio | At the end of training
  The waist circumference and hip circumference will be measured twice using an anthropometric tape while the participants stand erect and relaxed with their arms at their sides and feet positioned close together. The waist circumference will be measured between the upper border of the iliac crest and the lowest border of the rib cage at the end of normal expiration. The hip circumference will be measured at the widest part of the hip at the level of the greatest trochanter. The tape will be positioned at a level that is parallel to the floor. The unit of measure will be in centimeters (cm) to the nearest 0.1 cm. The waist-to-hip ratio will be calculated as the ratio of the waist-to-hip circumference.
Stroop Color-Word Test | One week before pretest
  Inhibition will be measured using the non-computerized Stroop Color and Word Test (under the word condition, color condition, and color-word condition in three separate 1-minute rounds. In the word condition (W), participants are instructed to read the Chinese words and name the Chinese colors printed in black. In the color condition (C), participants are required to name the colors of printed patches. Finally, in the color-word condition (CW), the name of a color (e.g., BLUE) is presented using either a congruent color (e.g., blue) or an incongruent color (e.g., yellow) in Chinese. Participants have to name the color, instead of reading the word as quickly and accurately as possible.
Stroop Color-Word Test | 10 weeks after intervention
  Inhibition will be measured using the non-computerized Stroop Color and Word Test (under the word condition, color condition, and color-word condition in three separate 1-minute rounds. In the word condition (W), participants are instructed to read the Chinese words and name the Chinese colors printed in black. In the color condition (C), participants are required to name the colors of printed patches. Finally, in the color-word condition (CW), the name of a color (e.g., BLUE) is presented using either a congruent color (e.g., blue) or an incongruent color (e.g., yellow) in Chinese. Participants have to name the color, instead of reading the word as quickly and accurately as possible.
Stroop Color-Word Test | 3 months after intervention
  Inhibition will be measured using the non-computerized Stroop Color and Word Test (under the word condition, color condition, and color-word condition in three separate 1-minute rounds. In the word condition (W), participants are instructed to read the Chinese words and name the Chinese colors printed in black. In the color condition (C), participants are required to name the colors of printed patches. Finally, in the color-word condition (CW), the name of a color (e.g., BLUE) is presented using either a congruent color (e.g., blue) or an incongruent color (e.g., yellow) in Chinese. Participants have to name the color, instead of reading the word as quickly and accurately as possible.
Digit Span Test | One week before pretest
  Working memory will be measured using the Backward Digit Span subtest of the Wechsler Intelligence Scale for Children, Third Edition [WISC-III]. Participants are orally presented with 18 sequences of single-digit numbers of increasing length, from two to nine (two sequences per length), and must repeat the numbers in backwards order. One point is given for each completely recalled sequence, and the test is terminated after two consecutive unsuccessful recalls.
Digit Span Test | 10 weeks after intervention
  Working memory will be measured using the Backward Digit Span subtest of the Wechsler Intelligence Scale for Children, Third Edition [WISC-III]. Participants are orally presented with 18 sequences of single-digit numbers of increasing length, from two to nine (two sequences per length), and must repeat the numbers in backwards order. One point is given for each completely recalled sequence, and the test is terminated after two consecutive unsuccessful recalls.
Digit Span Test | 3 months after intervention
  Working memory will be measured using the Backward Digit Span subtest of the Wechsler Intelligence Scale for Children, Third Edition [WISC-III]. Participants are orally presented with 18 sequences of single-digit numbers of increasing length, from two to nine (two sequences per length), and must repeat the numbers in backwards order. One point is given for each completely recalled sequence, and the test is terminated after two consecutive unsuccessful recalls.
Wisconsin Card Sorting Test | One week before pretest
  The Wisconsin Card Sorting Test will be administered with Inquisit 6 by Millisecond Software to measure cognitive flexibility. Participants are presented with four stimulus cards and a deck of response cards that vary in three dimensions (i.e., color, shape, and number). They are asked to match a fifth card from the sequentially presented response cards to one of the four key cards. The rules that underpin the classification are matching by color, shape, or number. Participants need to follow the correct card classification rule in accordance with the feedback they receive after each trial. After participants correctly respond to ten consecutive trials, the classification rule changes, requiring flexible set-shifting.
Wisconsin Card Sorting Test | 10 weeks after intervention
  The Wisconsin Card Sorting Test will be administered with Inquisit 6 by Millisecond Software to measure cognitive flexibility. Participants are presented with four stimulus cards and a deck of response cards that vary in three dimensions (i.e., color, shape, and number). They are asked to match a fifth card from the sequentially presented response cards to one of the four key cards. The rules that underpin the classification are matching by color, shape, or number. Participants need to follow the correct card classification rule in accordance with the feedback they receive after each trial. After participants correctly respond to ten consecutive trials, the classification rule changes, requiring flexible set-shifting.
Wisconsin Card Sorting Test | 3 months after intervention
  The Wisconsin Card Sorting Test will be administered with Inquisit 6 by Millisecond Software to measure cognitive flexibility. Participants are presented with four stimulus cards and a deck of response cards that vary in three dimensions (i.e., color, shape, and number). They are asked to match a fifth card from the sequentially presented response cards to one of the four key cards. The rules that underpin the classification are matching by color, shape, or number. Participants need to follow the correct card classification rule in accordance with the feedback they receive after each trial. After participants correctly respond to ten consecutive trials, the classification rule changes, requiring flexible set-shifting.

CONTACTS AND LOCATIONS:
Locations (1):
- The Education University of Hong Kong, Tai Po, Hong Kong

REFERENCES:
- [Derived] Poon K. Effects of Aerobic Exercise and High-Intensity Interval Training on the Mental Health of Adolescents Living in Poverty: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2022 Jan 17;11(1):e34915. doi: 10.2196/34915. PMID 35037892